CLINICAL TRIAL: NCT06983873
Title: Impact on Care Pathways of a New Management of Cervical Trauma in Conscious Patients Stable in Pre-hospital Care
Brief Title: IPSTRAUC : Impact on Care Pathways of a New Management of Cervical Trauma in Conscious Patients Stable in Pre-hospital Care
Acronym: IPSTRAUC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 35RC22_8872_IPSTRAUC; 2024-A00636-41 (Other: ID-RCB)
Record Dates: First submitted 2025-05-06; First posted 2025-05-21 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Prehospital Emergency; Neck Injury; Neck Trauma; Emergency Medical Services
MeSH Terms: conditions — Neck Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CCRa (Experimental): Pre-hospital management follow the rules of CCRa for all patients included in all sites ranodmized in the CCRa arm
  Interventions: Behavioral: adapted Canadian C-Spine rules
- Control (No Intervention): Patients included from all sites randomized in the control arm will be assessed according to standard practice

INTERVENTIONS:
Behavioral: adapted Canadian C-Spine rules — The CCRa are decision rules for pre-hospital cervical spine collar immobilization. They include three high-risk criteria indicating imaging, 5 low-risk criteria allowing assessment of cervical spine rotation, and finally the ability of patients to achieve limited active rotation. They have been designed and validated to avoid immobilization during transport to the emergency department without any significant cervical injury being missed.
  Arms: CCRa

SUMMARY:
The aim of the study is to evaluate the application of Canadian C-Spine rules adapted to pre-hospital settings in France in order to improve the appropriateness of cervical spine immobilisation, reduce unnecessary imaging examinations and optimise patient care pathways.

DETAILED DESCRIPTION:
The aim of this study is to assess the feasibility and effectiveness of applying the Canadian C-Spine rules adapted (CCRa) to the pre-hospital context of the French healthcare system. The hypothesis is that the use of these rules will improve the appropriateness of cervical collar use, reduce the need for imaging examinations, reduce referrals to emergency departments and ensure the identification of patients really at risk of cervical spine injury. Collaboration between primary care providers, including the fire service, emergency medical services (EMS) and general practitioners, will be crucial to successful implementation.

As part of routine care, each time the fire brigade is called out to deal with a health problem, it carries out an assessment at the SAMU (emergency medical service) to decide how the patient should be referred and treated. During this assessment and call, patients meeting the inclusion criteria of our study will be selected. After inclusion, patients will be assessed by a firefighter or SMUR physician specifically trained in CCRa rules in addition to the study training. Following application of the CCRa rules, the final decision on immobilisation will be taken by an investigating physician from the EMS in consultation with the study-trained professional taking charge of the patient. If the CCRa accept the indication for a cervical collar, immobilisation will be performed and the patient will be referred to the emergency department of the investigating centre. When the decision rules do not include an indication for cervical imaging, the patient will not be immobilised with a cervical collar. In this second case, patients will not be referred to A&E unless they have another reason for being referred to A&E. All patients included in the study will be recalled 14 and 30 days after their trauma to collect data about their healthcare consumption. At day 14, answers to a questionnaire focusing on cervical lesion suspicion are also collected. If there is a suspicion of a lesion in the answers to the questionnaire , the patient will be called in by the investigating centre for a medical examination and more detailed imaging tests. In parallel, the practices and organizations of firefighters in the fire stations will be evaluated before the start of inclusions and the feasibility and reproducibility of implementing CCRa as part of the pre-hospital care organisation of the French healthcare system will be determined.

ELIGIBILITY:
Inclusion Criteria:

PATIENTS

* GCS 15
* Stable (no organ failure, SBP ≥ 90 mmHg, DBP ≥ 65 mmHg, RF between 10 and 24 cycles/min)
* Cooperative (calm and obedient to instructions)
* Victim of a closed cervical spine trauma treated in the pre-hospital setting (fire brigade and/or Mobile Emergency and Resuscitation Service (SMUR)).
* Recent trauma (< 48 hours).
* Care regulated by the Emergency Medical Service (SAMU).
* Beneficiary of a social security scheme.
* Who can be contacted by telephone
* Have received oral and written information and have not objected to taking part in the study.

PROFESSIONAL

* Age ≥ 18 years
* Professional firefighter or EMS regulating doctor
* Professional who has received training in the protocol and, in the case of the experimental group, in the CCRa rules
* Fluency in French
* Having received oral and written information and not having objected to their participation in the study.

Exclusion Criteria:

PATIENTS

* Life-threatening organ damage
* Cardiorespiratory arrest since the traumatic event in question
* Polytrauma patient
* Penetrating trauma or a supra-clavicular wound following a knife or firearm injury
* Known spinal disease or previous spinal surgery (ankylosing spondylitis, rheumatic fever, spinal stenosis, cervical spine surgery).
* Acute paralysis (paraplegia, tetraplegia, hemiplegia, hemiparesis or documented sensory or motor deficit)
* Diagnosed osteogenesis imperfecta.
* Patients not regulated by EMS or transported to a hospital not participating in the study
* Pregnant or breast-feeding women
* Known situation of deprivation of liberty (safeguard of justice), guardianship or curatorship

PROFESSIONALS

- Persons referred to in articles L. 1121-5 to L. 1121-8 and L. 1122-1-2 of the Public Health Code (e.g. minors, protected adults, persons deprived of their liberty, persons under guardianship, curatorship, etc.).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 840 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2029-01 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients admitted to emergency service | Day 1
  Proportion of patients admitted to emergency following pre-hospital management of the traumatic event.

SECONDARY OUTCOMES:
Proportion of patients with cervical spine trauma admitted to emergency departments for a reason other than cervical spine trauma | Day 1
  Proportion of patients with cervical spine trauma admitted to emergency departments for a reason other than cervical spine trauma: Upper limb trauma, lower limb trauma, head trauma, chest pain, abdominal pain, pelvic pain, suture wound.
Rate of relevant management strategy | 14 days
  number of collars fitted and not fitted in a relevant manner in relation to the number of patients included in each of the two groups compared at day 14
Proportion of patients with cervical imagery at 14 days | 14 days
  Proportion of patients having undergone :
  - at least one cervical imaging within 14 days of the trauma (cervical X-rays, cervical CT or cervical MRI) and number of examinations carried out.
Proportion of patients with at least one consultation for neck pain | 30 days
  Proportion of patients having had at least one consultation for neck pain in the 30 days following the trauma (general practitioner in town or visit to the emergency department), number of consultations per patient and delay in relation to the initial treatment.
Cost of patient care | 30 days
  Cost of patient care at D30 from the point of view of the French National Health Insurance (transport, medical and paramedical consultations, cervical imaging, emergency room visits, hospitalisation).
ulcer complication rate of cervical collar immobilisation | Day 1
  - Percentage of patients with redness at the point of cervical collar compression compatible with an early stage of stage 1 pressure ulcer according to the National Pressure Ulcer Advisory Panel's classification of the different stages.
Overview of practices and organizations of firefighters in fire stations | 18 months
  Benefits and difficulties perceived in the adoption of new practices by teams of first-aiders and emergency medical service regulators
Proportion of patients with cervical imagery at 30 days | 30 days
  Proportion of patients having undergone :
  - at least one cervical imaging within 30 days of the trauma (cervical X-rays, cervical scanner or cervical MRI) and number of examinations performed
pain-linked complication rate of cervical collar immobilisation | Day 1
  - Assessment of pain in patients before and after fitting the cervical collar, using the Numerical Pain Scale (NPS): the NPS ranges from 0 to 10 (0 = no pain, 10 = unbearable pain).
Number of trained firefighters in fire stations | 18 months
  Percentage of professionals trained in the fire stations of the experimental group

CONTACTS AND LOCATIONS:
Overall Officials: François Saget, Md, Principal Investigator — CHU Rennes / Rennes University Hospital
Locations (12):
- France (12):
  - CHU Amiens-Picardie, Amiens
  - CHRU Besançon, Besançon
  - Centre Hospitalier Sud-Francilien, Corbeil-Essonnes
  - Hôpitaux La Rochelle Ré Aunis, La Rochelle
  - AP-HM Timone, Marseille
  - CHRU Nancy, Nancy
  - CHU Nice, Nice
  - CHU Poitiers, Poitiers
  - CHU Reims, Reims
  - CHU Rennes, Rennes
  - CHU Toulouse, Toulouse
  - Centre hospitalier Bretagne Atlantique, Vannes